CLINICAL TRIAL: NCT01412749
Title: Transoral Endoscopic Surgery Trial (TEST): A Registry for Endoscopic Head and Neck Surgery (eHNS)
Brief Title: TEST: Registry for Endoscopic Head and Neck Surgery
Acronym: TEST
Status: Terminated | Type: Observational
Why Stopped: Low Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: DR11-0131
Record Dates: First submitted 2011-08-08; First posted 2011-08-09 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Head and Neck Cancer
Keywords: registry; database; eHNS; Endoscopic Head and Neck Surgery; Transoral Endoscopic Surgery Trial; TEST; melanoma; head and neck surgery
MeSH Terms: conditions — Head and Neck Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- eHNS Participant Registry: Participants diagnosed with head and neck cancer who are candidates for definitive surgical resection of the primary tumor and who are candidates for eHNS.

SUMMARY:
The goal of this data review research study is to create a registry database using information (data) collected from patients who have had Endoscopic Head and Neck Surgery (eHNS). Researchers want to use the registry database to learn more about short-term and long-term outcomes for patients who have eHNS.

1.1 Primary Objective: To develop a registry database of patients who have had eHNS.

1.2 Secondary Objective: To evaluate short-term oncologic parameters and functional outcomes, operative for patients undergoing eHNS performed at M.D. Anderson Cancer Center (MDACC).

1.3 Tertiary Objective: To collect data on long-term oncologic outcomes including local and distant failure and survival following eHNS.

DETAILED DESCRIPTION:
Information from medical records will be collected and entered into the registry database at M. D. Anderson Cancer Center for future research related to cancer.

The information collected from medical records will include, but is not limited to, medical history, sex, age, race, gender, type and stage of disease, type of treatment(s) you have received, radiology reports, surgical and pathological reports, the results of any test(s), treatment(s) and/or surgery performed.

This is a registry study evaluating endoscopic head and neck surgery. The data from the surgical resection will be descriptive. Comparisons will be made to non-robotic, open historical controls and patients treated with radiation therapy, based on literature reports.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with head and neck cancer who are candidates for definitive surgical resection of the primary tumor and who, in the opinion of the treating MDACC physician, are candidates for eHNS will be included
2. Medically fit for an endoscopic surgical resection by consensus of MDACC surgical oncology and anesthesia faculty (common best practice criteria).
3. Date of records anticipated to be reviewed would be from March 1, 2011 to June 30, 2013
4. Approximately 200 patients are expected to fit the criteria above in order to be eligible for prospective data collection and review.

Exclusion Criteria:

None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals diagnosed with head and neck cancer and are a candidate to have endoscopic head and neck surgery (eHNS) for definitive resection of the primary tumor.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
eHNS Registry | 3 years
  Registry database using information (data) collected from participants who have had eHNS.

CONTACTS AND LOCATIONS:
Overall Officials: Christ Holsinger, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org